CLINICAL TRIAL: NCT01650961
Title: The Effect of Palonosetron on the QTc Interval During Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YSJeon_palonosetron_QTc
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Anesthesia, General; Palonosetron
MeSH Terms: interventions — Palonosetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Palonosetron (Experimental): Intravenous administration of palonosetron 0.075 mg before the induction of general anesthesia
  Interventions: Drug: Palonosetron
- Control (Placebo Comparator): Intravenous administration of normal saline before the induction of general anesthesia
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Palonosetron — 0.075 mg IV as bolus before induction of general anesthesia
  Other Names: Aloxi
  Arms: Palonosetron
Drug: Normal saline — 2 ml normal saline as bolus before induction of general anesthesia
  Arms: Control

SUMMARY:
The purpose of this study is to assess the effects of palonosetron on corrected QT interval duration during and after general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Elective abdominal surgery under general anesthesia

Exclusion Criteria:

* Cardiac valvular disease
* Clinically significant arrhythmias including atrial fibrillation
* Anti-emetics within 24 hours before surgery
* Steroids within 1 week before surgery
* Cancer chemotherapy or radiotherapy within 4 weeks before surgery
* Diabetes mellitus
* Pregnancy
* Patients receives a QT-prolonging drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
corrected QT interval (QTc interval) | up to 90 minutes after induction of general anesthesia
  at 2, 10, 15, 30, 60, 90 minutes after induction of general anesthesia, up to 1 minute after tracheal intubation

SECONDARY OUTCOMES:
proportion of patients whose corrected QT interval (QTc interval) is more than 450 ms for male or 470 ms for female | up to 2 hours after induction of general anesthesia
corrected QT interval (QTc interval) at Postanesthetic care unit | up to 1 hour after arrival on postanesthetic care unit
Incidence of postoperative nausea and vomiting | for 24 hours after surgery
proportion of patients who have more than 500 ms of corrected QT interval (QTc interval) | up to 2 hours after induction of general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Lee HC, Jung YS, Lee J, Min JJ, Hong DM, Choi EK, Oh S, Jeon Y. Effect of palonosetron on the QTc interval in patients undergoing sevoflurane anaesthesia. Br J Anaesth. 2014 Mar;112(3):460-8. doi: 10.1093/bja/aet335. Epub 2013 Oct 14. PMID 24129597